CLINICAL TRIAL: NCT00283686
Title: HALT Progression of Polycystic Kidney Disease Study A
Acronym: HALT PKD A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Boehringer Ingelheim (Industry); Merck Sharp & Dohme LLC (Industry); Polycystic Kidney Disease Foundation (Other); University of Pittsburgh (Other); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HALT PKD A; U01DK062401 (NIH); U01DK082230 (NIH)
Record Dates: First submitted 2006-01-26; First posted 2006-01-30 (Estimated); Results first posted 2015-02-27 (Estimated); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Kidney, Polycystic
Keywords: polycystic kidney disease; polycystic; kidney; disease; adpkd; halt; pkd; blood pressure; bp; hypertension; renal; renin-angiotensin-aldosterone-system; RAAS
MeSH Terms: conditions — Polycystic Kidney Diseases; Disease; Polycystic Kidney, Autosomal Dominant; Familial paroxysmal dystonia; Hypertension | interventions — Lisinopril; Angiotensin-Converting Enzyme Inhibitors; Telmisartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Study A, Arm 1 (Active Comparator): Lisinopril + Telmisartan (ACE-I + ARB) and standard blood pressure control of 120-130/70-80 mm Hg
  Interventions: Drug: Lisinopril; Drug: Telmisartan; Other: Standard Blood Pressure Control
- Study A, Arm 2 (Active Comparator): Lisinopril + Telmisartan (ACE-I + ARB) and low blood pressure control of 95-110/60-75 mm Hg
  Interventions: Drug: Lisinopril; Drug: Telmisartan; Other: Low Blood Pressure Control
- Study A, Arm 3 (Placebo Comparator): Lisinopril + Placebo (ACE-I + Placebo) and standard blood pressure control of 120-130/70-80 mm Hg
  Interventions: Drug: Lisinopril; Drug: Placebo; Other: Standard Blood Pressure Control
- Study A, Arm 4 (Placebo Comparator): Lisinopril + Placebo (ACE-I + Placebo) and low blood pressure control of 95-110/60-75 mm Hg
  Interventions: Drug: Lisinopril; Drug: Placebo; Other: Low Blood Pressure Control

INTERVENTIONS:
Drug: Lisinopril — Lisinopril titrated to 5mg, 10mg, 20mg, 40mg
  Other Names: ACE-I; ACE; Ace-Inhibitor
Drug: Telmisartan — Telmisartan/Placebo titrated to 40mg and 80mg, as tolerated by participants
  Other Names: ARB
  Arms: Study A, Arm 1; Study A, Arm 2
Drug: Placebo — Telmisartan/Placebo titrated to 40mg and 80mg, as tolerated by participants
  Arms: Study A, Arm 3; Study A, Arm 4
Other: Standard Blood Pressure Control — Achieve standard blood pressure control of 120-130/70-80 mm Hg using step dosing specified in protocol of lisinopril, study drug, hydrochlorothiazide, metoprolol, or non-dihydropyridine and dihydropyridine calcium channel blockers (diltiazem), clonidine, minoxidil, hydralazine at the discretion of the investigator
  Other Names: blood pressure control
  Arms: Study A, Arm 1; Study A, Arm 3
Other: Low Blood Pressure Control — Achieve low blood pressure control of 95-110/60-75 mm Hg using step dosing specified in protocol of lisinopril, study drug, hydrochlorothiazide, metoprolol, or non-dihydropyridine and dihydropyridine calcium channel blockers (diltiazem), clonidine, minoxidil, hydralazine at the discretion of the investigator
  Other Names: blood pressure control
  Arms: Study A, Arm 2; Study A, Arm 4

SUMMARY:
The efficacy of interruption of the renin-angiotensin-aldosterone system (RAAS) on the progression of cystic disease and on the decline in renal function in autosomal dominant kidney disease (ADPKD) will be assessed in two multicenter randomized clinical trials targeting different levels of kidney function: 1) early disease defined by GFR >60 mL/min/1.73 m2 (Study A); and 2) moderately advanced disease defined by GFR 25-60 mL/min/1.73 m2 (Study B; NCT01885559). Participants will be recruited and enrolled, either to Study A or B, over the first three years. Participants enrolled in Study A will be followed for at least 5 years, while those enrolled in Study B will be followed for five-to-eight years, with the average length of follow-up being six and a half years. The two concurrent randomized clinical trials differ by eligibility criteria, interventions and outcomes to be studied.

DETAILED DESCRIPTION:
* Specific Aims of Study A

To study the efficacy of angiotensin-converting-enzyme inhibitor (ACE-I) and angiotensin-receptor blockade (ARB) combination therapy as compared to ACE-I monotherapy and usual vs. low blood pressure targets on the percent change in kidney volume in participants with preserved renal function (GFR >60 mL/min/1.73m2)and high-normal blood pressure or hypertension (>130/80 mm Hg).

* Hypotheses to be tested in Study A

In ADPKD individuals with hypertension or high-normal blood pressure and relatively preserved renal function (GFR >60 mL/min/1.73 m2), multi-level blockade of the RAAS using ACE-I/ARB combination therapy will delay progression of cystic disease as compared to ACE-I monotherapy, and a low blood pressure goal will delay progression as compared with standard control.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ADPKD.
* Age 15-49 (Study A); Age 18-64 (Study B).
* GFR >60 mL/min/1.73 m2 (Study A); GFR 25-60 mL/min/1.73 m2 (Study B).
* BP ≥130/80 or receiving treatment for hypertension.
* Informed Consent.

Exclusion Criteria:

* Pregnant/intention to become pregnant in 4-6 yrs.
* Documented renal vascular disease.
* Spot urine albumin-to-creatinine ratio of >0.5 (Study A) or ≥1.0 (Study B) and/or findings suggestive of kidney disease other than ADPKD.
* Diabetes requiring insulin or oral hypoglycemic agents / fasting serum glucose of >126 mg/dl / random non-fasting glucose of >200 mg/dl.
* Serum potassium >5.5 milliequivalent per liter (mEq/L) for participants currently on ACE-I or ARB; >5.0 mEq/L for participants not currently on ACE-I or ARB.
* History of angioneurotic edema or other absolute contraindication for ACE-I or ARB. Intolerable cough associated with ACE-I is defined as a cough developing within six months of initiation of ACE-I in the absence of other causes and resolving upon discontinuation of the ACE-I.
* Indication (other than hypertension) for β-blocker or calcium channel blocker therapy (e.g. angina, past myocardial infarction, arrhythmia), unless approved by the site principal investigator. (PI may choose to accept an individual who is on only a small dose of one of these agents and would otherwise be eligible.)
* Systemic illness necessitating nonsteroidal antiinflammatory drugs (NSAIDs), immunosuppressant or immunomodulatory medications.
* Systemic illness with renal involvement.
* Hospitalized for acute illness in past 2 months.
* Life expectancy <2 years.
* History of non-compliance.
* Unclipped cerebral aneurysm >7mm diameter.
* Creatine supplements within 3 months of screening visit.
* Congenital absence of a kidney (also total nephrectomy for Study B).
* Known allergy to sorbitol or sodium polystyrene sulfonate.
* Exclusions specific to magnetic resonance imaging (Study A).

Ages: 15 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 558 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Schrier, M.D., Study Chair — University of Colorado, Denver; Arlene Chapman, M.D., Principal Investigator — Emory University; Ronald Perrone, M.D., Principal Investigator — Tufts University-New England Medical Center; Vicente Torres, M.D., Principal Investigator — Mayo Clinic; Marva Moxey-Mims, M.D., Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); Charity G Moore, MS,PhD, Principal Investigator — University of Pittsburgh
Locations (7):
- United States (7):
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - Tufts University-New England Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic Foundation, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Data are available at the NIDDK Central Repository, https://repository.niddk.nih.gov/studies/halt-pkd/?query=halt%20pkd
URL: https://repository.niddk.nih.gov/studies/halt-pkd/?query=halt%20pkd

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] Heerspink HJL, Inker LA, Tighiouart H, Collier WH, Haaland B, Luo J, Appel GB, Chan TM, Estacio RO, Fervenza F, Floege J, Imai E, Jafar TH, Lewis JB, Kam-Tao Li P, Locatelli F, Maes BD, Perna A, Perrone RD, Praga M, Schena FP, Wanner C, Xie D, Greene T; on behalf of CKD-EPI CT. Change in Albuminuria and GFR Slope as Joint Surrogate End Points for Kidney Failure: Implications for Phase 2 Clinical Trials in CKD. J Am Soc Nephrol. 2023 Jun 1;34(6):955-968. doi: 10.1681/ASN.0000000000000117. Epub 2023 Mar 15. PMID 36918388
- [Derived] Kim K, Trott JF, Gao G, Chapman A, Weiss RH. Plasma metabolites and lipids associate with kidney function and kidney volume in hypertensive ADPKD patients early in the disease course. BMC Nephrol. 2019 Feb 25;20(1):66. doi: 10.1186/s12882-019-1249-6. PMID 30803434
- [Derived] Schrier RW, Abebe KZ, Perrone RD, Torres VE, Braun WE, Steinman TI, Winklhofer FT, Brosnahan G, Czarnecki PG, Hogan MC, Miskulin DC, Rahbari-Oskoui FF, Grantham JJ, Harris PC, Flessner MF, Bae KT, Moore CG, Chapman AB; HALT-PKD Trial Investigators. Blood pressure in early autosomal dominant polycystic kidney disease. N Engl J Med. 2014 Dec 11;371(24):2255-66. doi: 10.1056/NEJMoa1402685. Epub 2014 Nov 15. PMID 25399733
- [Derived] Hogan MC, Abebe K, Torres VE, Chapman AB, Bae KT, Tao C, Sun H, Perrone RD, Steinman TI, Braun W, Winklhofer FT, Miskulin DC, Rahbari-Oskoui F, Brosnahan G, Masoumi A, Karpov IO, Spillane S, Flessner M, Moore CG, Schrier RW. Liver involvement in early autosomal-dominant polycystic kidney disease. Clin Gastroenterol Hepatol. 2015 Jan;13(1):155-64.e6. doi: 10.1016/j.cgh.2014.07.051. Epub 2014 Aug 9. PMID 25111236
- [Derived] Torres VE, Chapman AB, Perrone RD, Bae KT, Abebe KZ, Bost JE, Miskulin DC, Steinman TI, Braun WE, Winklhofer FT, Hogan MC, Oskoui FR, Kelleher C, Masoumi A, Glockner J, Halin NJ, Martin DR, Remer E, Patel N, Pedrosa I, Wetzel LH, Thompson PA, Miller JP, Meyers CM, Schrier RW; HALT PKD Study Group. Analysis of baseline parameters in the HALT polycystic kidney disease trials. Kidney Int. 2012 Mar;81(6):577-85. doi: 10.1038/ki.2011.411. Epub 2011 Dec 28. PMID 22205355
- See also: Polycystic Kidney Disease Foundation Website — http://www.pkdcure.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at seven clinical sites between February 2006 and June 2009.
Groups:
- ACE-I/ARB and Standard BP: ACE-I + angiotensin-receptor blocker (ARB) and standard blood pressure control of 120-130/70-80 mm Hg
  Lisinopril and Telmisartan: Lisinopril titrated to 5mg, 10mg, 20mg, 40mg and telmisartan titrated to 40mg and 80mg, as tolerated by participants, to achieve standard blood pressure control of 120-130/70-80 mm Hg.
- ACE-I/ARB and Low BP: ACE-I + angiotensin-receptor blocker (ARB) and low blood pressure control of 95-110/60-75 mm Hg
  Lisinopril and Telmisartan: Lisinopril titrated to 5mg, 10mg, 20mg, 40mg and telmisartan titrated to 40mg and 80mg, as tolerated by participants, to achieve low blood pressure control of 95-110/60-75 mm Hg.
- ACE-I/Placebo and Standard BP: ACE-I + Placebo and standard blood pressure control of 120-130/70-80 mm Hg
  Lisinopril and Placebo: Lisinopril titrated to 5mg, 10mg, 20mg, 40mg and placebo titrated to 40mg and 80mg, as tolerated by participants, to achieve standard blood pressure control of 120-130/70-80 mm Hg.
- ACE-I/Placebo and Low BP: ACE-I + Placebo and low blood pressure control of 95-110/60-75 mm Hg
  Lisinopril and Placebo: Lisinopril titrated to 5mg, 10mg, 20mg, 40mg and placebo titrated to 40mg and 80mg, as tolerated by participants, to achieve low blood pressure control of 95-110/60-75 mm Hg.
Period: Overall Study
Arm/Group | ACE-I/ARB and Standard BP | ACE-I/ARB and Low BP | ACE-I/Placebo and Standard BP | ACE-I/Placebo and Low BP
Started | 140 | 133 | 144 | 141
Completed | 111 | 92 | 111 | 109
Not Completed | 29 | 41 | 33 | 32
Not completed — Death | 1 | 1 | 1 | 0
Not completed — Lost to Follow-up | 21 | 31 | 26 | 20
Not completed — Less than full participation | 7 | 9 | 6 | 12

BASELINE CHARACTERISTICS:
Groups:
- ACE-I/ARB and Standard BP: ACE-I + ARB and standard blood pressure control of 120-130/70-80 mm Hg
  Lisinopril and Telmisartan: Lisinopril titrated to 5mg, 10mg, 20mg, 40mg and telmisartan titrated to 40mg and 80mg, as tolerated by participants, to achieve standard blood pressure control of 120-130/70-80 mm Hg.
- ACE-I/ARB and Low BP: ACE-I + ARB and low blood pressure control of 95-110/60-75 mm Hg
  Lisinopril and Telmisartan: Lisinopril titrated to 5mg, 10mg, 20mg, 40mg and telmisartan titrated to 40mg and 80mg, as tolerated by participants, to achieve low blood pressure control of 95-110/60-75 mm Hg.
- Total: Total of all reporting groups
Arm/Group | ACE-I/ARB and Standard BP | ACE-I/ARB and Low BP | ACE-I/Placebo and Standard BP | ACE-I/Placebo and Low BP | Total
Number analyzed (Participants) | 140 | 133 | 144 | 141 | 558
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (8.3) | 37.1 (8.4) | 35.8 (8.6) | 36.8 (8.0) | 36.7 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 64 | 73 | 70 | 275
  Male | 72 | 69 | 71 | 71 | 283
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 2 | 2 | 5
  Asian | 1 | 1 | 2 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 2 | 3 | 5 | 14
  White | 127 | 128 | 131 | 131 | 517
  More than one race | 5 | 2 | 6 | 2 | 15
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 2
Age at Diagnosis of autosomal dominant polycystic kidney disease (ADPKD) [Mean (Standard Deviation); unit: years] | 27.2 (10.0) | 28.5 (10.0) | 27.0 (9.5) | 27.6 (10.4) | 27.6 (10.0)
Body Mass Index (kg/m2) [Mean (Standard Deviation); unit: kg/m2] | 27.4 (5.4) | 27.4 (5.1) | 27.3 (5.5) | 26.8 (4.8) | 27.2 (5.2)
Serum Creatinine (mg/dl) [Mean (Standard Deviation); unit: mg/dl] | 1.0 (0.3) | 1.0 (0.2) | 0.9 (0.2) | 1.0 (0.2) | 1.0 (0.2)
Chronic Kidney Disease Epidemiology Collaboration (CKD EPI) eGFR (ml/min/m2) [Mean (Standard Deviation); unit: ml/min/m2] | 88.5 (18.8) | 86.5 (19.3) | 92.9 (18.5) | 87.6 (17.2) | 88.9 (18.5)
PKD Genotype [Number; unit: participants]
  PKD1 | 103 | 87 | 101 | 91 | 382
  PKD2 | 15 | 27 | 19 | 23 | 84
  No Mutation Detected | 10 | 10 | 12 | 14 | 46
  No information | 12 | 9 | 12 | 13 | 46

OUTCOME MEASURES:

1. Primary Outcome: Study A: Percent Annual Change in Total Kidney Volume
Description: Annual percentage change in total kidney volume as assessed by abdominal magnetic resonance imaging (MRI) at baseline, 2 years, 4 years, and 5 years follow-up.
Time Frame: Baseline and 2-, 4- and 5-year follow-up
Population: Analyses were conducted on all participants who had at least one total kidney volume measurement using intention to treat.
Measure: Mean (95% Confidence Interval); unit: percentage of Total Kidney Volume
Groups:
- ACE-I + ARB: ACE-I plus ARB (Lisinopril plus telmisartan)
- ACE-I Alone: ACE-I monotherapy (lisinopril only)
- Low Blood Pressure Group: Targeted blood pressure was 95/60 to 110/75 mm Hg
- Standard Blood Pressure Group: Targeted blood pressure was 120/70 to 130/80 mm Hg
Arm/Group | ACE-I + ARB | ACE-I Alone | Low Blood Pressure Group | Standard Blood Pressure Group
Number analyzed (Participants) | 271 | 282 | 271 | 282
percentage of Total Kidney Volume | 6.0 [5.5 to 6.4] | 6.2 [5.7 to 6.7] | 5.6 [5.2 to 6.1] | 6.6 [6.1 to 7.1]
Statistical Analysis 1: Comparison: ACE-I + ARB vs ACE-I Alone; Test type: Superiority or Other; p = 0.52, Mixed Models Analysis — adjusted for age, sex, race, baseline estimated GFR, and clinical site; Test for differences between treatment groups over time; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.8 to 5.0]
Statistical Analysis 2: Comparison: Low Blood Pressure Group vs Standard Blood Pressure Group; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis — adjusted for age, sex, race, baseline estimated GFR, and clinical site; Testing differences between blood pressure groups over time; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-1.6 to -0.2]

2. Secondary Outcome: Kidney Function (eGFR)
Description: The estimated GFR was calculated by means of the Chronic Kidney Disease Epidemiology Collaboration equation with the use of central serum creatinine measurements.
Time Frame: Up to 96 months (6 month assessments)
Population: Analyses were intention to treat: All participants who were randomized.
Measure: Mean (95% Confidence Interval); unit: ml/min/1.73/m2/yr
Arm/Group | ACE-I + ARB | ACE-I Alone | Low Blood Pressure Group | Standard Blood Pressure Group
Number analyzed (Participants) | 273 | 284 | 274 | 283
ml/min/1.73/m2/yr | -3.0 [-3.3 to -2.7] | -2.9 [-3.2 to -2.6] | -2.9 [-3.2 to -2.6] | -3.0 [-3.3 to -2.7]
Statistical Analysis 1: Comparison: ACE-I + ARB vs ACE-I Alone; Test type: Superiority or Other; p = 0.52, Mixed Models Analysis — adjusting for age, sex, race, and clinical site; Testing for differences in treatment over time (differences in slopes over time); Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.6 to 0.3]
Statistical Analysis 2: Comparison: Low Blood Pressure Group vs Standard Blood Pressure Group; Test type: Superiority or Other; p = 0.55, Mixed Models Analysis — adjusted for age, sex, race, and clinical site; Testing for differences between groups over time (differences in slopes over time); Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.3 to 0.6]

3. Secondary Outcome: Albuminuria
Description: Urine albumin excretion, centrally processed from 24 hour urine collection
Time Frame: Up to 96 months (assessed annually)
Population: Analysis by intention to treat
Measure: Mean (95% Confidence Interval); unit: annual percent change in mg/24 hr
Arm/Group | ACE-I + ARB | ACE-I Alone | Low Blood Pressure Group | Standard Blood Pressure Group
Number analyzed (Participants) | 273 | 284 | 274 | 283
annual percent change in mg/24 hr | -1.1 [-3.1 to 0.8] | -0.4 [-2.3 to 1.6] | -3.8 [-5.7 to -1.8] | 2.4 [0.5 to 4.4]
Statistical Analysis 1: Comparison: ACE-I + ARB vs ACE-I Alone; Test type: Superiority or Other; p = 0.57, Mixed Models Analysis; adjusting for age, sex, race, and clinical site; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-3.3 to 1.9]
Statistical Analysis 2: Comparison: Low Blood Pressure Group vs Standard Blood Pressure Group; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; adjusting for age, sex, race, and clinical site; Mean Difference (Final Values) = -6.1, 95% CI 2-sided [-8.5 to -3.4]

4. Secondary Outcome: Aldosterone
Description: Urinary aldosterone excretion, centrally processed, 24 hour urine collection
Time Frame: Up to 96 months (assessed annually)
Population: Analysis using intention to treat
Measure: Mean (95% Confidence Interval); unit: annual % change micrograms per 24 hr
Arm/Group | ACE-I + ARB | ACE-I Alone | Low Blood Pressure Group | Standard Blood Pressure Group
Number analyzed (Participants) | 273 | 284 | 274 | 283
annual % change micrograms per 24 hr | -8.5 [-9.9 to -7.2] | -7.3 [-8.7 to -5.9] | -8.5 [-9.9 to -7.1] | -7.3 [-8.6 to -5.9]
Statistical Analysis 1: Comparison: ACE-I + ARB vs ACE-I Alone; Test type: Superiority or Other; p = 0.18, Mixed Models Analysis; adjusting for age, sex, race, and clinical site; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-3.1 to 0.6]
Statistical Analysis 2: Comparison: Low Blood Pressure Group vs Standard Blood Pressure Group; Test type: Superiority or Other; p = 0.19, Mixed Models Analysis; adjusting for age, sex, race, and clinical site; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-3.1 to 0.6]

5. Secondary Outcome: Left Ventricular Mass Index
Description: Left ventricular mass index (g/m^2) measured by MRI, centrally reviewed and measured
Time Frame: 0, 24 months, 48 months, 60 months
Population: Analyses were conducted using intention to treat for participants with at least one left ventricular mass index measure.
Measure: Mean (95% Confidence Interval); unit: annual change in g/m^2
Arm/Group | ACE-I + ARB | ACE-I Alone | Low Blood Pressure Group | Standard Blood Pressure Group
Number analyzed (Participants) | 268 | 274 | 265 | 277
annual change in g/m^2 | -0.91 [-1.15 to -0.68] | -0.83 [-1.06 to -0.59] | -1.17 [-1.41 to -0.93] | -0.57 [-0.80 to -0.34]
Statistical Analysis 1: Comparison: ACE-I + ARB vs ACE-I Alone; Test type: Superiority or Other; p = 0.58, Mixed Models Analysis; adjusted for age, sex, race, baseline estimated GFR, and clinical site; Mean Difference (Final Values) = -0.088, 95% CI 2-sided [-0.40 to 0.22] — comparing the annual change over time between ACE/ARB and ACE alone
Statistical Analysis 2: Comparison: Low Blood Pressure Group vs Standard Blood Pressure Group; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; adjusted for age, sex, race, baseline estimated GFR, and clinical site; Mean Difference (Net) = -0.60, 95% CI 2-sided [-0.91 to -0.29] — comparing annual change in LVMI between Low Blood Pressure and Standard Blood Pressure groups

6. Secondary Outcome: Renal Blood Flow
Description: renal blood flow (mL/min/1.73 m^2) from MRI, centrally reviewed and measured. This outcome was more difficult to measure resulting in more missing data than other MRI outcomes such as total kidney volume (TKV) and left ventricular mass index (LVMI).
Time Frame: 0, 24 months, 48 months, 60 months
Population: Analyses were conducted using intention to treat analyses for participants with at least one valid renal blood flow measure.
Measure: Mean (95% Confidence Interval); unit: annual change in mL/min/1.73 m^2
Arm/Group | ACE-I + ARB | ACE-I Alone | Low Blood Pressure Group | Standard Blood Pressure Group
Number analyzed (Participants) | 233 | 247 | 236 | 244
annual change in mL/min/1.73 m^2 | -6.6 [-11.0 to -2.1] | -9.5 [-14.0 to -5.1] | -7.6 [-12.0 to -3.1] | -8.5 [-13.0 to -4.1]
Statistical Analysis 1: Comparison: ACE-I + ARB vs ACE-I Alone; Test type: Superiority or Other; p = 0.29, Mixed Models Analysis; adjusted for age, sex, race, baseline estimated GFR, and clinical site; Mean Difference (Final Values) = 2.97, 95% CI 2-sided [-2.55 to 8.50] — difference in annual change in mL/min/1.73 m^2 for ACE+ARB compared to ACE alone
Statistical Analysis 2: Comparison: Low Blood Pressure Group vs Standard Blood Pressure Group; Test type: Superiority or Other; p = 0.73, Mixed Models Analysis; adjusting for age, sex, race, baseline estimated GFR, and clinical site; Mean Difference (Final Values) = 0.98, 95% CI 2-sided [-4.54 to 6.50] — difference in annual change mL/min/1.73 m^2 between low and standard blood pressure groups

7. Secondary Outcome: All-Cause Hospitalizations
Time Frame: Up to 96 months
Population: Intention to treat analysis: All participants who were randomized.
Measure: Number; unit: events
Arm/Group | ACE-I + ARB | ACE-I Alone | Low Blood Pressure Group | Standard Blood Pressure Group
Number analyzed (Participants) | 273 | 285 | 274 | 284
events | 85 | 128 | 93 | 120
Statistical Analysis 1: Comparison: ACE-I + ARB vs ACE-I Alone; Test type: Superiority or Other; p = 0.0228, Regression, Cox; adjusting for age, sex, race, and clinical site; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.53 to 0.95]
Statistical Analysis 2: Comparison: Low Blood Pressure Group vs Standard Blood Pressure Group; Test type: Superiority or Other; p = 0.59, Regression, Cox; adjusting for age, sex, race, and clinical site; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.70 to 1.22]

8. Secondary Outcome: Quality of Life Physical Component Summary
Description: Short Form-36 Quality of Life Physical Component Summary ranges from 0 (worst possible outcome) to 100 (best possible outcome)
Time Frame: baseline, 12, 24, 36, 48, 60, 72, 84, and 96 months (assessed annually)
Population: Analysis using intention to treat
Measure: Mean (95% Confidence Interval); unit: annual change in units on a scale
Arm/Group | ACE-I + ARB | ACE-I Alone | Low Blood Pressure Group | Standard Blood Pressure Group
Number analyzed (Participants) | 273 | 285 | 274 | 284
annual change in units on a scale | -0.24 [-0.37 to -0.11] | -.23 [-.35 to -0.10] | -0.17 [-0.30 to -0.03] | -0.30 [-0.43 to -0.17]
Statistical Analysis 1: Comparison: ACE-I + ARB vs ACE-I Alone; Test type: Superiority or Other; p = 0.87, Mixed Models Analysis; adjusting for age, sex, race, and clinical site; Mean Difference (Final Values) = -0.016, 95% CI 2-sided [-0.19 to 0.17]
Statistical Analysis 2: Comparison: Low Blood Pressure Group vs Standard Blood Pressure Group; Test type: Superiority or Other; p = 0.14, Mixed Models Analysis; adjusting for age, sex, race, and clinical site; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.046 to 0.31]

9. Secondary Outcome: Quality of Life Mental Component Summary
Description: Short Form-36 Quality of LIfe Mental Component Summary ranges from 0 (worst possible outcome) to 100 (best possible outcome)
Time Frame: baseline, 12, 24, 36, 48, 60, 72, 84, and 96 months (assessed annually)
Population: Analysis using intention to treat.
Measure: Mean (95% Confidence Interval); unit: annual change in units on a scale
Arm/Group | ACE-I + ARB | ACE-I Alone | Low Blood Pressure Group | Standard Blood Pressure Group
Number analyzed (Participants) | 273 | 285 | 274 | 284
annual change in units on a scale | 0.19 [0.03 to 0.35] | -0.06 [-0.21 to 0.10] | -0.05 [-0.21 to 0.11] | 0.18 [0.03 to 0.33]
Statistical Analysis 1: Comparison: ACE-I + ARB vs ACE-I Alone; Test type: Superiority or Other; p = 0.0221, Mixed Models Analysis; adjusting for age, sex, race, and clinical site; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [0.036 to 0.46]
Statistical Analysis 2: Comparison: Low Blood Pressure Group vs Standard Blood Pressure Group; Test type: Superiority or Other; p = 0.0339, Mixed Models Analysis; adjusting for age, sex, race, and clinical site; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.44 to -0.018]

ADVERSE EVENTS:
Time Frame: 5-8 years with average follow-up of 5.7 years
Arm/Group | ACE-I + ARB | ACE-I Alone | Low Blood Pressure Group | Standard Blood Pressure Group
Serious Adverse Events (participants affected / at risk) | 58/273 | 90/285 | 69/274 | 79/284
Other Adverse Events (participants affected / at risk) | 23/273 | 21/285 | 23/274 | 21/284
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACE-I + ARB (N=273) | ACE-I Alone (N=285) | Low Blood Pressure Group (N=274) | Standard Blood Pressure Group (N=284)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (3) | 3 (4) | 1 (1) | 3 (6)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Aortic valve disease (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 6 (9) | 3 (5) | 6 (7)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ileal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Death NOS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Pain (General disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (2)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 5 (5) | 2 (2) | 3 (3)
Appendicitis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hepatitis viral (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Joint infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ovarian infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 3 (3) | 2 (2)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4) | 4 (4) | 1 (1)
Akathisia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 4 (5) | 2 (2) | 3 (4)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pregnancy, puerperium and perinatal conditions - Other, specify (Pregnancy, puerperium and perinatal conditions) | 9 (11) | 11 (14) | 10 (13) | 10 (12)
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 7 (8) | 6 (7) | 9 (10) | 4 (5)
Renal calculi (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Renal colic (Renal and urinary disorders) | 2 (2) | 2 (2) | 0 (0) | 4 (4)
Renal hemorrhage (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Breast atrophy (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Uterine pain (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Uterine obstruction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 1 (2) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 7 (7) | 2 (2) | 5 (5)
Hypertension (Vascular disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (3)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACE-I + ARB (N=273) | ACE-I Alone (N=285) | Low Blood Pressure Group (N=274) | Standard Blood Pressure Group (N=284)
Acute kidney injury (Renal and urinary disorders) | 13 (15) | 16 (19) | 16 (17) | 13 (17)
Hyperkalemia (Metabolism and nutrition disorders) | 11 (13) | 5 (6) | 7 (8) | 9 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No